CLINICAL TRIAL: NCT03662308
Title: Developing a Feedback-Controlled Heated Vest to Address Thermoregulatory Dysfunction in Persons With Spinal Cord Injury
Brief Title: Heated Vest for Persons With Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: United States Military Academy West Point (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: B2884-P; 1I21RX002884-01A1 (NIH)
Record Dates: First submitted 2018-07-30; First posted 2018-09-07 (Actual); Results first posted 2024-02-01 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Spinal Cord Injuries
Keywords: Hypothermia; Body Temperature Regulation; Cognition
MeSH Terms: conditions — Spinal Cord Injuries; Hypothermia

STUDY DESIGN:
Intervention Model Description: After the heated vest has 1) been fully bench-tested and 2) satisfied safety and tolerability testing in able-bodied subjects, it will be tested in persons with tetraplegia using a crossover design with the order of the two visits randomized.
  1. Thermal Challenge with heated vest (subjects with tetraplegia only): Subjects with tetraplegia, while seated and wearing only a standard T-shirt and shorts, will be fitted with an appropriately sized heated vest. Subjects will be transferred to a pre-cooled thermal chamber and data will be collected for up to 2 hours with the self-regulating heated vest.
  2. Thermal Challenge with non-heated vest (subjects with tetraplegia only): The same subjects with tetraplegia (from Visit 2), while seated and wearing only a standard T-shirt and shorts, will be fitted with an appropriately sized, similar, but non-heated vest. Subjects will be transferred to a pre-cooled thermal chamber and data will be collected for up to 2 hours.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Heated Vest Safety & Comfort (able-bodied subjects) (Other): Able-bodied controls will be fitted with an appropriately sized heated vest, while wearing only a standard cotton T-shirt and shorts, and will remain seated in a wheelchair. Subjects will be transferred to a pre-cooled (18 degrees C) thermal chamber and data will be collected for 2 hours with the heated vest on full power. Outcome Variables for Visit 1: Skin thermocouple temperatures, subjective ratings of thermal sensation.
  Interventions: Device: Heated Vest
- Heated Vest Efficacy (persons with tetraplegia) (Experimental): Subjects with tetraplegia, while seated and wearing only a standard cotton T-shirt and shorts, will be fitted with an appropriately sized heated vest. Subjects will be transferred to a pre-cooled (18 degrees C) thermal chamber and data will be collected for up to 2 hours with the self-regulating heated vest. Primary Dependent variables: core body temperature (Tcore), cognitive performance, and thermal comfort.
  Interventions: Device: Heated Vest
- Non-Heated Vest control condition (persons with tetraplegia) (Active Comparator): The same subjects with tetraplegia from the experimental arm, while seated and wearing only a standard cotton T-shirt and shorts, will be fitted with an appropriately sized, similarly insulated, but non-heated vest (control condition). Subjects will be transferred to a pre-cooled (18 degrees C) thermal chamber and data will be collected for up to 2 hours with the non-heated vest. Primary Dependent variables: core body temperature (Tcore), cognitive performance, and thermal comfort.
  Interventions: Device: Non-Heated Vest

INTERVENTIONS:
Device: Heated Vest — Heated vest that regulates its heat output based on the user's skin, the user's core temperature, and the ambient temperature
  Other Names: Feedback-controlled heated vest
  Arms: Heated Vest Efficacy (persons with tetraplegia); Heated Vest Safety & Comfort (able-bodied subjects)
Device: Non-Heated Vest — A similarly insulated (compared to the experimental vest), but non-heated vest
  Other Names: Active comparator vest, control condition
  Arms: Non-Heated Vest control condition (persons with tetraplegia)

SUMMARY:
Persons with higher levels of spinal cord injury (above the 2nd thoracic vertebrae; tetraplegia) are unable to maintain normal core body temperature (Tcore) when exposed to cool environments. In persons with tetraplegia, even limited exposure to cool temperatures may cause Tcore to approach hypothermic values and impair cognitive performance. Conversely, an increase in Tcore from subnormal to normal range may improve cognitive performance. Prior work has shown that cool seasonal temperatures have an adverse effect on personal comfort and the ability to perform vital daily activities of self-care in persons with tetraplegia. Interventions that address the vulnerability to hypothermia are limited. A self-regulating heated vest designed specifically for persons with tetraplegia is a novel and promising strategy to address this problem. By more effectively maintaining Tcore, the vest can decrease the adverse impact of cool temperatures on comfort, quality of life, and performance of vital daily tasks for Veterans with tetraplegia during the cooler seasons.

DETAILED DESCRIPTION:
Persons with spinal cord injury (SCI), particularly cervical injuries (tetraplegia), are unable to effectively regulate core body temperature (Tcore) due to interruption of motor, sensory, and sympathetic pathways. Thus, control of distal extremity vasoconstriction (heat conservation) and shivering thermogenesis (heat production) are impaired, and the ability to maintain a constant Tcore is compromised. Persons with tetraplegia often report "feeling cold," frequently present with subnormal Tcore (35-36.5 degrees C), and are particularly vulnerable to hypothermia (Tcore<35 degrees C) and associated impairment in cognitive performance, even when exposed to temperatures that are comfortable for able-bodied (AB) individuals. Cool seasonal temperatures have been shown to have a greater adverse effect on personal comfort, activities of daily living (ADLs), and vital daily activities in persons with tetraplegia than that of AB controls. Conversely, a minimal increase in Tcore from subnormal to normothermia, secondary to ambient heat may improve cognitive performance. Interventions addressing the tendency to poikilothermia and enhanced vulnerability to hypothermia in persons with tetraplegia are limited. Therefore, exploration of safe and efficacious bioengineering solutions to address the physiological, cognitive, and quality of life (QoL) issues associated with the routine exposure to cool temperatures that persons with tetraplegia often encounter is warranted.

The goals of this pilot study are to: 1) fully bench-test the heated vest for safety before performing any human subject testing; 2) study the safety and tolerability of a feedback-controlled heated vest in AB controls; and 3) study the efficacy of this heated vest to minimize the expected decline in Tcore and associated deterioration of cognitive performance during 2 hours of cool exposure in persons with tetraplegia.

In persons with tetraplegia, a two-condition (heated vest, non-heated vest) prospective study is being proposed to compare the physiological and cognitive responses to 2 hours of controlled cool exposure (18 degrees C) with a prototype heated vest vs. a similar, but non-heated vest (control condition). Eight subjects with tetraplegia (C3-T1, AIS A and B) and eight AB controls will be recruited for study participation. Before the prototype is tested on human subjects, it will have been fully bench tested and have satisfied all safety requirements and specifications. AB subjects will be observed to ensure the safety of the vest, which will be accomplished by determining the temperatures of the vest ( 39 degrees C) and subjective thermal sensation of no greater than "warm" during a cool condition that will be identical to the condition which subjects with SCI will be exposed. Subjects with tetraplegia will test the efficacy of the heated vest, i.e. preventing the expected decline in Tcore and cognitive performance and increase in thermal comfort.

After the feedback-controlled heated vest has been fully bench-tested and has satisfied all safety requirements (interior vest temperature does not exceed 39 degrees C at maximal power) and design specifications (lightweight, slim, easy to don doff), the following specific aims will be addressed:

Primary Specific Aim: In a cool thermal chamber (18 degrees C), AB controls will wear the heated vest at maximal setting for 120 minutes in the seated position to determine (1) maximum temperatures of all areas of the interior (user's side) of the heated vest and (2) subjective comfort of the heated vest (safety testing).

Primary Hypotheses: The study of AB controls will demonstrate (1) All areas under the vest will have temperatures 39 degrees C. (2) All subjects will report a thermal sensation no greater than "warm" this would include identification of "hot spots" (Zhang 9-point Thermal Sensation Scale).

Secondary Specific Aim: During exposure to a cool environment (18 degrees C) for up to 120 minutes in the seated position, persons with tetraplegia will wear the heated vest to determine (1) change in Tcore, (2) change in cognitive performance, and (3) change in thermal comfort (efficacy testing).

Secondary Hypotheses: In persons with tetraplegia wearing the heated vest compared to the same persons wearing the non-heated vest, it's expected that (1) 30% of the subjects will have a decline of 0.5 degrees C in Tcore compared with 80% in the control condition, (2) 30% of the subjects will demonstrate a decline of at least 1 T-score in at least one of the following measures: Interference of Stroop Color and Word test, Digit Span of Wechsler Adult Intelligence Scale-Fourth Edition, compared with 80% in the control condition, and (3) a greater percentage of subjects reporting increased thermal comfort (Zhang 6-point Comfort Scale).

ELIGIBILITY:
Inclusion Criteria:

Subjects with spinal cord injury (SCI) and able-bodied subjects will be recruited according to the following criteria:

* Duration of injury 1 year
* Neurological Level of SCI [C3-T1]; American Spinal Injury Association (ASIA) Impairment Scale (AIS) A & B
* Euhydration

  * Subjects will be instructed to avoid caffeine and alcohol
  * maintain normal salt and water intake
  * avoid strenuous exercise for 24 hours prior to study

Exclusion Criteria:

* Known heart, kidney, peripheral vascular or cerebrovascular disease
* High blood pressure
* History of Traumatic Brain Injury (TBI) or diagnosed cognitive impairment
* Untreated thyroid disease
* Diabetes mellitus
* Acute illness or infection
* Dehydration
* Smoking
* Pregnant women
* BMI>30 kg/m2
* Broken, inflamed, or otherwise fragile skin

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-02-25 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Philip Handrakis, PT DPT EdD, Principal Investigator — James J. Peters Veterans Affairs Medical Center
Locations (1):
- James J. Peters VA Medical Center, Bronx, NY, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang H, Huizenga C, Arens E, Wang D. Thermal sensation and comfort in transient non-uniform thermal environments. Eur J Appl Physiol. 2004 Sep;92(6):728-33. doi: 10.1007/s00421-004-1137-y. PMID 15221406
- See also: Spinal Cord Damage Research Center — http://www.scirc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Persons With Tetraplegia: Heated Vest First, Then Non-Heated Vest: Subjects with tetraplegia, while seated and wearing only a standard cotton T-shirt and shorts, will be fitted with an appropriately sized heated vest. Subjects will be transferred to a pre-cooled (18 degrees C) thermal chamber and data will be collected for up to 2 hours with the self-regulating heated vest. Primary Dependent variables: core body temperature (Tcore), cognitive performance, and thermal comfort.
  Then, the same subjects with tetraplegia from the experimental arm, while seated and wearing only a standard cotton T-shirt and shorts, will be fitted with an appropriately sized, similarly insulated, but non-heated vest (control condition). Subjects will be transferred to a pre-cooled (18 degrees C) thermal chamber and data will be collected for up to 2 hours with the non-heated vest. Primary Dependent variables: core body temperature (Tcore), cognitive performance, and thermal comfort.
- Persons With Tetraplegia: Non-Heated Vest First, Then Heated Vest: Subjects with tetraplegia, while seated and wearing only a standard cotton T-shirt and shorts, will be fitted with an appropriately sized, insulated, but non-heated vest (control condition). Subjects will be transferred to a pre-cooled (18 degrees C) thermal chamber and data will be collected for up to 2 hours with the non-heated vest. Primary Dependent variables: core body temperature (Tcore), cognitive performance, and thermal comfort.
  Then, the same subjects with tetraplegia from the experimental arm, while seated and wearing only a standard cotton T-shirt and shorts, will be fitted with an appropriately sized heated vest. Subjects will be transferred to a pre-cooled (18 degrees C) thermal chamber and data will be collected for up to 2 hours with the self-regulating heated vest. Primary Dependent variables: core body temperature (Tcore), cognitive performance, and thermal comfort.
Period: First Intervention
Arm/Group | Heated Vest Safety & Comfort (Able-bodied Subjects) | Persons With Tetraplegia: Heated Vest First, Then Non-Heated Vest | Persons With Tetraplegia: Non-Heated Vest First, Then Heated Vest
Started | 8 | 5 | 4
Completed | 8 | 5 | 4
Not Completed | 0 | 0 | 0
Period: Second Intervention (Tetraplegia ONLY)
Arm/Group | Heated Vest Safety & Comfort (Able-bodied Subjects) | Persons With Tetraplegia: Heated Vest First, Then Non-Heated Vest | Persons With Tetraplegia: Non-Heated Vest First, Then Heated Vest
Started | 0 | 5 | 4
Completed | 0 | 5 | 4
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase 2: Persons With Tetraplegia: For Persons with Tetraplegia: Heated Vest First, then Non-Heated Vest
  Subjects with tetraplegia, while seated and wearing only a standard cotton T-shirt and shorts, will be fitted with an appropriately sized heated vest. Subjects will be transferred to a pre-cooled (18 degrees C) thermal chamber and data will be collected for up to 2 hours with the self-regulating heated vest. Primary Dependent variables: core body temperature (Tcore), cognitive performance, and thermal comfort.
  Then, the same subjects with tetraplegia from the experimental arm, while seated and wearing only a standard cotton T-shirt and shorts, will be fitted with an appropriately sized, similarly insulated, but non-heated vest (control condition). Subjects will be transferred to a pre-cooled (18 degrees C) thermal chamber and data will be collected for up to 2 hours with the non-heated vest. Primary Dependent variables: core body temperature (Tcore), cognitive performance, and thermal comfort.
  For Persons with Tetraplegia: Non-Heated Vest First, then Heated Vest
  The subjects underwent the same interventions, but in the opposite order. That is, subjects with tetraplegia, while seated and wearing only a standard cotton T-shirt and shorts, will be fitted with an appropriately sized insulated, but non-heated vest (control condition), then with a an appropriately sized insulated, heated vest.
- Total: Total of all reporting groups
Arm/Group | Heated Vest Safety & Comfort (Able-bodied Subjects) | Phase 2: Persons With Tetraplegia | Total
Number analyzed (Participants) | 8 | 9 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 8 | 15
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.5 (14.6) | 44.33 (14) | 42.06 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 6 | 8 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 7 | 8 | 15
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 9 | 17
BMI [Mean (Standard Deviation); unit: kg/(m^2)] | 23.96 (2.8) | 26.30 (3.2) | 25.2 (3.3)

OUTCOME MEASURES:

1. Primary Outcome: Change in Core Body Temperature (Tcore)
Description: Tcore will be continuously monitored throughout baseline and thermal challenge periods (with heated & non-heated vests) by a TX-2 Rectal probe and Iso-Thermex Multichannel Thermometer (Columbus Instruments, Columbus, OH). The probe will be placed 10 cm beyond the anal sphincter.
Time Frame: Visits 2 & 3 (subjects with tetraplegia only): Continuously throughout baseline & Thermal Challenge (2 hrs) periods. The change in Tcore from baseline to the end of Thermal Challenge will be determined.
Population: Tcore measurement was not performed in able-bodied participants.
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Heated Vest Safety & Comfort (Able-bodied Subjects) | Heated Vest Efficacy (Persons With Tetraplegia) | Non-Heated Vest Control Condition (Persons With Tetraplegia)
Number analyzed (Participants) | 0 | 9 | 9
Degrees Celsius |  | -0.22 (.34) | -0.46 (0.24)
Statistical Analysis 1: Comparison: Heated Vest Efficacy (Persons With Tetraplegia) vs Non-Heated Vest Control Condition (Persons With Tetraplegia); Test type: Superiority; p < 0.05, ANOVA; Mean Difference (Final Values) = .6

2. Primary Outcome: Change in Cognitive Performance: WAIS-IV (Wechsler Adult Intelligence Scale-Fourth Edition)
Description: WAIS-IV Digit Span test has 3, 16-point sections (Forward, Backward, Sequence) and assesses attention, processing speed, and working memory.
  Cognitive battery is administered at BL, after Thermal Challenge (tetra only). Testing conditions are distraction-free.
  The Forward section has 16 numerical sequences of successive increasing length (each 1 point). Participant is read the numbers, then asked to repeat the test numbers in the same order. In Backward, participant is asked to repeat the numbers in reverse order. In Sequence portion, the participant is asked to repeat the numbers in ascending order.
  Sections add to a WAIS-IV Total Score of 48. The greater the score, the better the cognitive function. The minimum score, which would represent not being able to repeat even the first sequence of numbers, is 0.
  We report the difference in WAIS-IV score before and after the cold challenge. The more negative the difference, the more cognitive impairment after cold challenge.
Time Frame: Visits 2 & 3 (subjects with tetraplegia only): At the end baseline (at 15 min) & end of Thermal Challenge (at 120 min) periods. The change in cognitive performance from baseline to the end of Thermal Challenge will be determined. Each WAIS is 10 min
Population: We did not administer the Wechsler Adult Intelligence Scale Test to able-bodied participants.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Heated Vest Safety & Comfort (Able-bodied Subjects) | Heated Vest Efficacy (Persons With Tetraplegia) | Non-Heated Vest Control Condition (Persons With Tetraplegia)
Number analyzed (Participants) | 0 | 9 | 9
score on a scale |  | -0.500 (0.707) | -0.375 (0.460)

3. Primary Outcome: Change in Cognitive Performance: Delayed Recall
Description: Delayed Recall section of the Montreal Cognitive Assessment (MoCA): Subjects will be asked to repeat 5 simple words immediately and then recall them after a 5-minute delay to assess working memory.
  In scoring the MoCA, one point is awarded for each of the five words. Thus, the score ranges from 0 (no words remembered) to 5 (all words remembered). A higher score represents a more intact delayed recall capacity.
  We administered the Delayed Recall of the MoCA before and after the cold challenge, in both the heated vest (powered) and non-heated vest control condition. The reported measure is the mean difference in MoCA Delayed Recall scores before and after the cold challenge. Here, a more negative number represents a greater degree of impairment in delayed recall (working memory) after the cold challenge.
Time Frame: Visits 2 & 3 tetraplegia only): At the end baseline (at 15 min) & end of Thermal Challenge (at 120 min) periods. The change in cognitive performance from baseline to the end of Thermal Challenge will be determined. Each assessment requires 6 min.
Population: We did not measure working memory in able bodied participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Heated Vest Safety & Comfort (Able-bodied Subjects) | Heated Vest Efficacy (Persons With Tetraplegia) | Non-Heated Vest Control Condition (Persons With Tetraplegia)
Number analyzed (Participants) | 0 | 9 | 9
score on a scale |  | -0.38 (0.74) | -2.00 (1.8)

4. Primary Outcome: Change in Cognitive Performance: Stroop
Description: Stroop Color and Word: Subjects will be asked to read words of colors, colors of fonts to assess attention and processing speed; color of fonts of words which describe conflicting colors to assess response inhibition (executive functioning).
  Each assessment is 4 min.
  The Stroop Test yields three scores. The Raw Word score is the number of words correctly completed on the Word page in 45 seconds. Similarly for Color, and Color-Word. For example, in the color-word section, a participant correctly identifying the color of 61 words, the score is 61.
  Greater scores reflects greater executive functioning. Zero is the minimum score, which corresponds to not being able to read any of the words of colors or colors of fonts. Each words of colors or color of fonts correctly identified in time confer 1 point.
  We report the difference in Word-Color before the cold challenge and after the cold challenge, for each intervention. Negative differences represent impaired executive function.
Time Frame: Visits 2 & 3 (subjects with tetraplegia only): At the end baseline (at 15 min) & end of Thermal Challenge (at 120 min) periods. The change in cognitive performance from baseline to the end of Thermal Challenge will be determined.
Population: We did not measure cognitive performance in able bodied participants.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Heated Vest Safety & Comfort (Able-bodied Subjects) | Heated Vest Efficacy (Persons With Tetraplegia) | Non-Heated Vest Control Condition (Persons With Tetraplegia)
Number analyzed (Participants) | 0 | 9 | 9
score on a scale |  | -2.125 (1.302) | -1.750 (1.590)

5. Secondary Outcome: Change in Thermal Comfort (TC)
Description: Thermal Comfort will be measured every 10 minutes throughout BL and thermal challenge periods by the Zhang 6-point thermal comfort scale: +3 (very comfortable), +2 (comfortable), +1 (just comfortable), -1 (just uncomfortable), -2 (uncomfortable), and -3 (very uncomfortable). A greater frequency of +1, +2, and +3 scores are considered more desirable than -1, -2, and -3 scores during the Thermal Challenge.
  Each assessment requires only the time needed for the subject to respond (typically less than 10 seconds).
Time Frame: Visits 1, 2, & 3 (all subjects): During baseline & every 10 minutes throughout Thermal Challenge (2 hrs). The change in TC from baseline to the end of Thermal Challenge will be determined.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Heated Vest Safety & Comfort (Able-bodied Subjects) | Heated Vest Efficacy (Persons With Tetraplegia) | Non-Heated Vest Control Condition (Persons With Tetraplegia)
Number analyzed (Participants) | 8 | 9 | 9
score on a scale | 0.031 (.72) | -1.04 (1.51) | -0.96 (1.12)

6. Other Pre Specified Outcome: Change in Skin Temperature (Tsk) Under the Heated Vest
Description: Skin thermocouples (TX-4 Skin Surface probes, Columbus Instruments, Columbus, OH) will be taped to 12 sites on the anterior trunk. Tsk data will be collected continuously throughout the baseline (BL) and Thermal Challenge periods. All areas under the vest will have skin temperatures less than or equal to 39 degrees C.
Time Frame: Visits 2 & 3 (all subjects): Continuously throughout baseline (15 min) & Thermal Challenge (2 hrs) periods. The change in Tsk from baseline to the end of Thermal Challenge will be determined.
Measure: Mean (Standard Deviation); unit: Degrees Celcius
Arm/Group | Heated Vest Safety & Comfort (Able-bodied Subjects) | Heated Vest Efficacy (Persons With Tetraplegia) | Non-Heated Vest Control Condition (Persons With Tetraplegia)
Number analyzed (Participants) | 8 | 9 | 9
Degrees Celcius | 3.79 (1.26) | 4.64 (1.20) | 0.77 (0.42)

7. Other Pre Specified Outcome: Change in Thermal Sensation (TS)
Description: Thermal sensation will be measured on the Zhang 9-point Thermal Sensation scale: +4 (very hot), +3 (hot), +2 (warm), +1 (slightly warm), 0 (neutral), -1 (slightly cool), -2 (cool), -3 (cold), and -4 (very cold). TS should be no greater than "warm" this would include identification of "hot spots".
  Each assessment requires only the time needed for the subject to respond (typically less than 10 seconds).
Time Frame: Visit 1 (able-bodied subjects only): During baseline & every 10 minutes throughout Thermal Challenge (2 hrs). The change in TS from baseline to the end of Thermal Challenge will be determined.
Population: We did not collect Thermal Sensation in persons with tetraplegia; we only collected this outcome measure in able-bodied controls.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Heated Vest Safety & Comfort (Able-bodied Subjects) | Heated Vest Efficacy (Persons With Tetraplegia) | Non-Heated Vest Control Condition (Persons With Tetraplegia)
Number analyzed (Participants) | 8 | 0 | 0
units on a scale | 0.59 (0.61) |  |

ADVERSE EVENTS:
Time Frame: Data was collected during the duration of the study (one day for able-bodied participants, and approximately two weeks, as scheduling allowed, for individuals with cervical spinal cord injuries).
Description: The definition used is that on clinical trials.
Arm/Group | Heated Vest Safety & Comfort (Able-bodied Subjects) | Heated Vest Efficacy (Persons With Tetraplegia) | Non-Heated Vest Control Condition (Persons With Tetraplegia)
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/8 | 0/9 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-25): https://cdn.clinicaltrials.gov/large-docs/08/NCT03662308/Prot_SAP_000.pdf